CLINICAL TRIAL: NCT04961905
Title: A Phase I Clinical Trial to Compare and Evaluate the Pharmacokinetic Characteristics and Safety After Administration of NVP-2002 and Co-administration of NVP-2002-R1 and NVP-2002-R2 in Healthy Adult Volunteers
Brief Title: Pharmacokinetic Characteristics and Safety After Administration of NVP-2002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NVP Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NVP-2002_BA
Record Dates: First submitted 2021-06-29; First posted 2021-07-14 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single tablet fist, fasted (Experimental): single tablets of NVP-2002-R1 and NVP-2002-R2 followed by NVP-2002 FDC, fasted condition
  Interventions: Drug: NVP-2002-R1+NVP-2002-R2
- FDC fist, fasted (Experimental): NVP-2002 FDC followed by single tablets of NVP-2002-R1 and NVP-2002-R2, fasted condition
  Interventions: Drug: NVP-2002
- Single tablet fist, fed (Experimental): single tablets of NVP-2002-R1 and NVP-2002-R2 followed by NVP-2002 FDC, fasted condition
  Interventions: Drug: NVP-2002-R1+NVP-2002-R2
- FDC fist, fed (Experimental): NVP-2002 FDC followed by single tablets of NVP-2002-R1 and NVP-2002-R2, fasted condition
  Interventions: Drug: NVP-2002

INTERVENTIONS:
Drug: NVP-2002-R1+NVP-2002-R2 — NVP-2002-R1 1 tablet, once daily and NVP-2002-R2 1 tablet, once daily
  Arms: Single tablet fist, fasted; Single tablet fist, fed
Drug: NVP-2002 — NVP-2002 is a combination of NVP-2002-R1 and NVP-2002_R2 NVP-2002, 1 tablet, once daily
  Arms: FDC fist, fasted; FDC fist, fed

SUMMARY:
The purpose of this study is to compare and evaluate the pharmacokinetic characteristics and safety after administration of NVP-2002 and co-administration of NVP-2002-R1 and NVP-2002-R2 in healthy adult volunteers.

DETAILED DESCRIPTION:
Phase 1 to evaluate the pharmacokinetic characteristics and safety after administration of NVP-2002 and co-administration of NVP-2002-R1 and NVP-2002-R2. Which is designed as ramdomized, oral, single dose, 2×2 crossover.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult subjects who signed informed consent
* Body Mass Index(BMI)=18.5~29.9kg/㎡

Exclusion Criteria:

* Subjects participated in another clinical trial within 6 months prior to administration of the study drug
* Inadequate subject for the clinical trial by the investigator's decision
* Upper Limits of Normal x 1.5 < Aspartate transaminase(AST), Alanine transminase(ALT), Total bilirubin

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-09-03 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of plasma: Cmax | 0hours - 72hours
  Cmax of NVP-2002-R1 and NVP-2002-R2
Pharmacokinetics of plasma: AUCt | 0hours - 72hours
  Area under the curve of NVP-2002-R1 and NVP-2002-R2

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, M.D., Ph.D, Principal Investigator — Jeonbuk National University Hospital
Locations (1):
- Jeonbuk national university hospital, Jeonju, Jeollabuk-do, South Korea